CLINICAL TRIAL: NCT02235038
Title: A Mechanistic Examination of Dietary Composition on Metabolic Fuels Availability
Brief Title: Metabolic Fuels Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Framingham State University (Other); Brigham and Women's Hospital (Other); Boston Medical Center (Other); Nutrition Science Initiative (Other); New Balance Foundation (Other)
Responsible Party: Principal Investigator, David S. Ludwig, MD, PhD, Director, Obesity Prevention Center, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB-P00014678
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet, Carbohydrate-Restricted; Carbohydrates; CD36 Antigens; Proteins; Diet, High-Protein Low-Carbohydrate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low carbohydrate diet (Active Comparator)
  Interventions: Behavioral: Low carbohydrate diet
- Moderate carbohydrate diet (Active Comparator)
  Interventions: Behavioral: Moderate carbohydrate diet
- High carbohydrate diet (Active Comparator)
  Interventions: Behavioral: High carbohydrate diet

INTERVENTIONS:
Behavioral: Low carbohydrate diet — Composition (by proportion of calories) : 15% carbohydrate, 65% fat, 20% protein
  Other Names: Composition : 15% carbohydrate, 65% fat, 20% protein
  Arms: Low carbohydrate diet
Behavioral: Moderate carbohydrate diet — Feeding study. Composition (by proportion of calories): 40% carbohydrate, 40% fat, 20% protein
  Arms: Moderate carbohydrate diet
Behavioral: High carbohydrate diet — Feeding study. Composition (by proportion of calories): 60% carbohydrate, 20% fat, 20% protein
  Arms: High carbohydrate diet

SUMMARY:
This study will evaluate a potential physiologic mechanism underlying the effects of dietary composition on control of body weight

DETAILED DESCRIPTION:
The challenge in maintaining long-term weight loss is well known, however new research suggests diet quality may be the driving factor. A pilot study from our group demonstrated that a higher carbohydrate-containing diet was associated with lower total energy expenditure during weight loss maintenance (Ebbeling et al). These findings will be confirmed in the ongoing Framingham State Food Study (NCT02068885): Following weight loss on a standard diet, 150 overweight or obese adults (aged 18 to 65 years) will be randomized to one of three weight-loss maintenance diets varying in carbohydrate to fat ratios for 20 weeks.

However, the specific mechanisms underlying the calorie-independent effects of diet remain unclear. Another study from our group demonstrated lower energy availability (calculated based on caloric content of circulating metabolic fuel concentrations) in the fasting and late post-prandial periods in 8 overweight or obese young adults who were maintained on a low-fat (high-carbohydrate) diet (Walsh et al). We hypothesize that this lower metabolic fuel availability on a high carbohydrate diet results in part from increased anabolic changes within the adipocyte, favoring fat storage in preference to oxidation.

We will invite subjects already enrolled in the Framingham State Food Study to participate, aiming for a total of 30 subjects (with the goal of approximately equal numbers per diet group following randomization to assigned test diet in the parent study). Participants will be admitted to a research unit for a 24-hour period during weight maintenance on the test diet, during which they will undergo frequent blood sampling for the measurement of circulating metabolic fuels, hunger and satiety ratings, while consuming their assigned diet meals. Each participant will also undergo two abdominal subcutaneous fat aspiration biopsies under local anesthesia, the first immediately following weight loss (before initiating the test diet) and the second during weight maintenance, in order to perform gene expression analyses on the adipose tissue. Our main outcomes will be a comparison in energy availability (the sum of energy in the major metabolic fuels in the blood) between diet groups in the late postprandial period and changes in adipose tissue gene expression within-individuals and by diet group assignment. Other outcomes will include differences in hunger and satiety ratings, total 24-hour energy availability, and specific metabolic fuel concentrations.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria (as detailed in Framingham State Food Study, NCT02068885)

* Aged 18 to 65 years
* BMI ≥ 25 kg/m2
* BMI < 40 kg/m2 and weight ≤ 300 lbs (136 kg)
* Medical clearance from a primary care provider
* Student or employee at Framingham State University throughout enrollment in the study
* Willing and able to eat and drink only the foods and beverages on the study menus
* Willing to eat in the dining hall
* Willing to abstain from consuming alcohol during participation

Additional Inclusion Criteria:

• Willing to undergo additional procedures in this ancillary study

Exclusion Criteria:

Exclusion Criteria (as detailed in Framingham State Food Study, NCT02068885)

* Change in body weight exceeding ±10% during prior year
* Recent adherence to a special diet
* Recent adherence to a vigorous physical activity regimen (e.g., participation in a varsity sport)
* Chronic use of any medication or dietary supplement that could affect study outcomes
* Current smoking (1 cigarette in the last week)
* Heavy baseline alcohol consumption or history of binge drinking
* Physician diagnosis of a major medical/psychiatric illness or eating disorder
* Abnormal blood glucose, TSH, CBC, BUN, Creatinine
* ALT greater than 150% of the normal upper limit
* Plans for a vacation during the study that would preclude adherence to prescribed diet
* Additional exclusions for female participants: Irregular menstrual cycles; any change in birth control medication during the 3 months prior to enrollment; pregnancy or lactation during the 12 months prior to enrollment

Additional Exclusion Criteria:

* Allergy or prior reaction to Lidocaine
* Medical condition or medication that would increase risk of bleeding, infection or skin reactions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2016-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Late postprandial energy availability | 10 - 15 weeks after initiation of test diets
  Post-prandial energy availability calculated as the sum, in kcal/L, of energy from circulating metabolic fuels (glucose, non-esterified fatty acids, lactate and ketoacids), as measured during a 24 hr inpatient admission. Time of interest includes 2.5 - 5 hr in the postprandial period after breakfast, lunch and dinner.

SECONDARY OUTCOMES:
Late postprandial energy availability, with lactate excluded | 10 - 15 weeks after initiation of test diets
  Post-prandial energy availability calculated as the sum, in kcal/L, of energy from circulating metabolic fuels (glucose, non-esterified fatty acids, and ketoacids), as measured during a 24 hr inpatient admission. Time of interest includes 2.5 - 5 hr in the postprandial period after breakfast, lunch and dinner. (Lactate is metabolized primarily by the liver, which uses this substrate to produce glucose. Thus, including lactate in the calculation of metabolic fuels may comprise "double counting" -- and not accurately reflect actual fuel availability to body tissues)
Fasting energy availability | 10 - 15 weeks after initiation of test diet
  Fasting energy availability calculated as the sum, in kcal/L, of energy from circulating metabolic fuels (glucose, non-esterified fatty acids, lactate and ketoacids), as measured during a 24 hr inpatient admission.
Total energy availability | 10 - 15 weeks after initiation of test diets
  Total energy availability calculated as the sum, in kcal/L, of energy from circulating metabolic fuels (glucose, non-esterified fatty acids, lactate and ketoacids), as measured during a 24 hr inpatient admission.
Hunger | 10 - 15 weeks after initiation of test diets
  Measured during a 24 hr inpatient admission.
Satiety | 10 - 15 weeks after initiation of test diets
  Measured during a 24 hr inpatient admission.
Glucose | 10 - 15 weeks after initiation of test diets
  Concentration during 24-hr inpatient admission
Non-esterified fatty acids | 10 - 15 weeks after initiation after test diet
  Concentration during 24-hr inpatient admission
Lactate | 10 - 15 weeks after initiation of test diets
  Concentration during 24-hr inpatient admission
Ketoacids | 10 - 15 weeks after initiation of test diets
  Concentration during 24-hr inpatient admission
Insulin | 10 - 15 weeks after initiation of test diets
  Concentration during 24-hr inpatient admission

OTHER OUTCOMES:
Effect modification by insulin secretion | 10 - 15 weeks after initiation of test diets
  We will test for an interaction by insulin secretion (as measured by plasma insulin 30 minutes into a standard oral glucose tolerance test) of the relationship between diet and metabolic fuels concentration.
Adipocyte studies of anabolic status | 10 - 15 weeks after initiation of test diets
  Adipose tissue gene expression studies (assessed by mRNA levels of selected candidate genes involved in lipid storage, fatty acid and lipid biosynthesis, angiogenesis, inflammation). Change from baseline.
Adipose tissue histology | 10 - 15 weeks after initiation of test diets
  Change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Shams, MD, Study Director — Boston Children's Hospital; David s Ludwig, MD, PhD, Principal Investigator — Boston Children's Hospital; Cara B Ebbeling, PhD, Principal Investigator — Boston Children's Hospital
Locations (4):
- United States (4):
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Framingham State University, Framingham, Massachusetts

REFERENCES:
- [Background] Walsh CO, Ebbeling CB, Swain JF, Markowitz RL, Feldman HA, Ludwig DS. Effects of diet composition on postprandial energy availability during weight loss maintenance. PLoS One. 2013;8(3):e58172. doi: 10.1371/journal.pone.0058172. Epub 2013 Mar 6. PMID 23483989
- [Background] Ebbeling CB, Swain JF, Feldman HA, Wong WW, Hachey DL, Garcia-Lago E, Ludwig DS. Effects of dietary composition on energy expenditure during weight-loss maintenance. JAMA. 2012 Jun 27;307(24):2627-34. doi: 10.1001/jama.2012.6607. PMID 22735432